CLINICAL TRIAL: NCT06250842
Title: Assessing the Cognitive Effects of Chronic Benzodiazepine Use in Patients: A Comprehensive Study Using fNIRs and PET/MRI Technologies
Brief Title: Benzodiazepine Impact on Cognitive Function: fNIRs and PET/MRI Study
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PJ-KS-KY-2023-577
Record Dates: First submitted 2024-01-26; First posted 2024-02-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-02

CONDITIONS: Benzodiazepine Adverse Reaction; Depression, Anxiety; Benzodiazepine Dependence
Keywords: Benzodiazepines; Long Term Adverse Effects; Cognitive Neuroscience; Neuroendocrinology; immunomodulatory potential
MeSH Terms: conditions — Depression; Anxiety Disorders; Long Term Adverse Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Long-term benzodiazepine use group: Continuous use of benzodiazepines for ≥3 months
- Non-benzodiazepine use group: No history of prior benzodiazepine use
- Healthy Controls: Healthy Controls

SUMMARY:
This study explores the impact of long-term benzodiazepine (BZDs) use on cognitive function and associated neuroimaging markers. While BZDs are established treatments for conditions like anxiety and insomnia, recent warnings highlight risks, including neurocognitive effects. Neuroimaging studies indicate potential neuroprotective effects of BZDs. Functional near-infrared spectroscopy (fNIRS) measures cerebral cortex function during cognitive tasks. Combining fNIRS with mood and cognitive scales, this study assesses cortical activation. 2-deoxy-2-fluoro-D-glucose-positron emission tomography (FDG-PET) evaluates brain metabolism. DPA-714 PET assesses neuroinflammation. The primary objective is to compare brain functional activation, metabolism, and neuroinflammatory levels between long-term BZD users and non-users. This comprehensive approach aims to provide insights into BZD effects on cognition and associated brain markers.

DETAILED DESCRIPTION:
Benzodiazepines(BZDs) have been long-established treatments for various conditions, including anxiety disorders and insomnia. Recent FDA warnings emphasize the risks of misuse and dependence associated with BZDs. Epidemiological investigations have consistently raised concerns regarding the long-term utilization of GABAergic medications, such as BZD and Z-drugs, due to their observed association with an elevated likelihood of neurocognitive impairments, including the development of Alzheimer's disease(AD). Recent neuroimaging studies have provided insights into the neuroprotective effects of BZD. These studies reveal that prolonged use of BZD in humans is associated with reduced amyloid deposition and a greater hippocampus volume. Functional near-infrared spectroscopic imaging utilizes changes in measured near-infrared light to monitor relative changes in oxyhemoglobin and deoxyhemoglobin concentrations in the cerebral cortex, allowing the detection of dynamic changes in cerebral cortical function during cognitive processing states. In this study, investigators will use functional near-infrared spectroscopy (fNIRS) to measure oxygenated (HbO2), deoxygenated hemoglobin (HbR), and total hemoglobin activation in various parts of the cortex, combined with mood and cognitive scales.

Brain metabolism, measured using 2-deoxy-2-fluoro-D-glucose-positron emission tomography (FDG-PET) imaging, can guide clinicians in both research and clinical evaluation, with specific patterns of brain metabolism reduction aiding in the diagnosis of AD or related disorders. The PET tracer DPA-714, binding to the 18 kDa translocator protein (TSPO), provides a non-invasive measure of neuroinflammation in activated microglia/macrophages within the mitochondria. The primary objective of this study is to observe differences in brain functional activation, brain metabolism, and brain neuroinflammatory levels between subjects on long-term BZDs use and those not taking BZDs.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous use of benzodiazepines for ≥3 months, matched with participants who have not taken benzodiazepines.
2. Education time ≥6 years.
3. Abstained from alcohol, coffee, and other psychoactive substances in the 24 hours before the examination.

Exclusion Criteria：

1. Brain damage due to various reasons (such as head trauma, dementia, epilepsy, brain tumors, etc.).
2. Severe systemic diseases (such as malignant tumors, etc.).
3. Acute cerebrovascular disease in the past 3 months. History of substance abuse other than benzodiazepines (such as alcohol, opioids, etc.).
4. Inability to cooperate with fNIRS, PET/MRI examinations, and scale assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The First Affiliated Hospital of Dalian Medical University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-11 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Brain hemodynamic activity with fNIRS | for 3 years
  This includes changes in the concentration of oxygenated and deoxygenated hemoglobin as measured by the change in light absorption, along with comprehensive analyses of activation values and functional connectivity.
Longitudinal evolution of biomarkers measured from neuroimaging (including structural, functional, and multimodal MRI) and molecular neuroimaging (18F-FDG PET/MRI、DPA-714-PET/MRI) | for 3 years
  Estimates of brain TSPO concentrations measured with PET will serve as a marker for neuroinflammation. Variation of the regional cerebral glucose consumption and TSPO-PET measures, derived from neuroimaging (including structural, functional, and multimodal MRI), will be compared between three groups.

SECONDARY OUTCOMES:
Mini-Mental State Evaluation (MMSE) | About 15 min during the study visit
  Clinician-administered screening tool used to systematically and thoroughly assess mental status through five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. Scores range between 0-30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Scores of Hamilton Depression Scale | About 15 min during the study visit
  Using to assess depressive symptoms. With higher scores associated with more severe depression symptoms. Total scores <7 is normal; Mild depression with total scores of 7～17; Moderate depression with total scores of 18～24; Total scores >24 for severe depression.
Scores of Hamilton Anxiety Scale | About 15 min during the study visit
  Using to assess anxiety symptoms. With higher scores associated with more severe anxiety symptoms. Total scores< 7 indicates no anxiety; Total scores≥7 indicates possible anxiety; Total scores≥14 indicates anxiety; Total scores≥21 indicates obvious anxiety; Total scores≥29 points indicates serious anxiety.
Pittsburgh Sleep Quality Index | About 15 min during the study visit
  Using to assess the sleep quality. Total scores of 0-5 indicates that the quality of sleep is very good, 6～10 indicates that the quality of sleep is OK, 11～15 indicates that the quality of sleep is average, and 16～21 indicates that the quality of sleep is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Hui min Zhang, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China